CLINICAL TRIAL: NCT04819763
Title: Training of the Lateral Pterygoid Muscle in the Treatment of Anterior Temporomandibular Joint Disc Displacement With Reduction With Pain
Brief Title: Physical Exercises for Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0016032021
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Facial Pain; Temporomandibular Disorder; Temporomandibular Joint Disorders; Temporomandibular; Functional Disturbance
Keywords: physical therapy; stabilization appliance; clinical trial; dentistry
MeSH Terms: conditions — Facial Pain; Temporomandibular Joint Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Prospective, randomized study with control group, stratified by gender.
Who Masked: Outcomes Assessor
Masking Description: Unblinded with respect to the examiner and to the patient, blinded to the statisticians in the evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical training of the lateral pterygoid muscle (Experimental): Static stretching and isometric contraction exercises of the lateral pterygoid muscle are used to strengthen and restore a physiological lateral movement of the mandible.
  Interventions: Other: Physical therapy
- Stabilization appliance therapy (Active Comparator): Hard acrylic splint with anterior canine guidance for the lower jaw.
  Interventions: Other: Appliance therapy

INTERVENTIONS:
Other: Physical therapy — Coordination training for lateral movement of the mandible (spatula exercise):
  1. A wooden spatula is loosely placed between the teeth of the upper and lower jaw; the head must be aligned with the body axis; the exercise should be performed in front of a mirror.
  2. The lower jaw moves to the left and back to the center with little contact to the spatula
  3. The lower jaw moves to the right and back to the center under contact with the spatula
  Training of the left lateral pterygoid muscle:
  1. The left palm is placed on the left temple region
  2. Right hand forms a fist and is placed on the tip of the right chin
  3. Both arms are aligned parallel to the surface of the floor
  4. The lower jaw is moved to the right against a moderate resistance of the fist = concentric muscle work
  5. With measured force of the fist, the lower jaw is brought back to the center = eccentric muscle work (Right lateral pterygoid muscle training with opposite hands.)
  Arms: Physical training of the lateral pterygoid muscle
Other: Appliance therapy — Upper and lower jaw impressions are registered by using an intraoral scanner. The arbitrary hinge axis position is determined using a face bow.
  The stabilization appliance with anterior canine guidance is manufactured in the Lexmann laboratory in Dresden.
  The stabilization appliance is incorporated by the dentist and the static and dynamic occlusion is checked. A tension-free fit of the appliance on the lower jaw is necessary. Additionally, equal contacts in the side teeth area and incisors guidance in the case of mandibular protrusion are checked visually and by using occlusion foil. During mandibular lateral movement only the canine guidance takes place and is also registered optically and by using occlusion foil.Interference contacts should be adjusted.
  The patient is instructed to wear the stabilization appliance while sleeping. The wearing rhythm is described as intermittent. (three nights - wearing the appliance, one night - not wearing the appliance).
  Arms: Stabilization appliance therapy

SUMMARY:
Temporomandibular Disorders are a common clinical picture that appear in particular in people between the age of 20 and 40 years. About 33% of the total population shows symptoms and signs of TMD. Among the temporomandibular joint disorders anterior disc displacement appear to be the most common. In case of limitations of jaw movements and or pain conservative methods including combinations of behavior change, physiotherapy, stabilization appliance therapy and medication are most popular. The benefit of a self-treatment program to strengthen the lateral pterygoid muscle and to learn a properly executed lower jaw sideways movement to achieve pain reduction is up to now not well investigated. The aim of this study is to examine the effectiveness of muscle training for the treatment of patients with anterior disc displacement with reduction (DDWR). 60 patients with DDWR and pain (≥18 years) will be randomly allocated to two groups: 1. Physical exercises, 2. Stabilization appliance therapy. All patients receive a functional examination according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) at baseline.

The training in group 1 includes eccentric and concentric counter-movements of the lower jaw muscle to strengthen and restore a physiological lateral movement of the mandible. The muscle exercises should be performed once a day with 5-6 repetitions per side. The treatment with an equilibration appliance in the lower jaw serves as a comparison group. Patients are instructed to wear the appliance while sleeping. The wearing rhythm is described as intermittent. (three nights - wearing the appliance, one night - not wearing the appliance). The primary target variable is the occurrence of pain in the head and joint area before and during therapy. The variable is measured using a numeric rating scale (NRS; 0-10) during the baseline examination and control check-ups after 2, 4 and 6 months.

DETAILED DESCRIPTION:
The literature describes the cause of a temporomandibular disorder (TMD) as a multifactorial event. It can be influenced by anatomical, neuromuscular, traumatic or psychosocial factors. Disturbances often occur in the condyle-disc complex of the temporomandibular joint. The relationship between the articular disc and the condyle head is pathologically altered. The Diagnostic Criteria for Temporomandibular disorders (DC / TMD) describe the displacement of the disc in 4 different forms: disc displacement with reduction; disc displacement with reduction and intermittent locking; disc displacement without reduction with limited opening and disc displacement without reduction without limited opening. TMDs are a common clinical picture that appears in particular in people between the age of 20 and 40 years. About 33% of the total population show signs and symptoms of TMD.

Studies prove that the displacement of the disc with reduction is the most common disorder among temporomandibular joint disorders. According to the DC / TMD, this clinical picture shows intracapsular and biomechanical alterations. If the mouth is closed, the articular disc is often located in front of the mandibular condyle; if the mouth is opened, the disc moves back to its original position on the condyle. Anterior disc displacement appears to be the most common, although a medial or lateral displacement is also possible. During the disc repositioning clicking, popping or snapping noises are usually recorded. Temporomandibular joint disorders such as disc displacement, can also cause pain. Overstretching of the posterior ligament and a compression of the bilaminar zone mandibular movements can be pain-related. Therefore, clicking, popping or snapping noises in the area of the temporomandibular joint (TMJ) correlate with pain in the surrounding tissue. Those complaints intensify when opening the mouth or chewing food.

The treatment of TMD should be oriented on evidence-based procedures that are easy to implement in practice and have a long-term positive effect on the patient's symptoms. Conservative methods including combinations of behavior change, physiotherapy, splint-therapy and medication are most popular. The physiotherapeutic treatment should pursue different strategies, including manual therapy methods (e.g. mobilization and stretching of the temporomandibular joint and / or the neck area) and the demonstration of exercises in everyday life (e.g. self-mobilization and stretching of the masticatory muscles and / or cervical spine) and in addition educating the patient (e.g. about the perception of parafunctions or relaxation techniques). Conservative attempts for patients with TMD should be the first choice. However, there is still no clear data situation and the data pool of randomized clinical studies on this topic needs to be improved. So far studies demonstrate a positive effect of the tested therapy forms. But the individual studies differ greatly in terms of the patient pool, diagnosis, treatment modalities and the result. Furthermore, a precisely described procedure is missing in some papers. Therefore, an exact reproducibility for practitioners is not executable. More research is needed into the benefits of various non-invasive treatments for TMD.

The primary goal of this study is to decrease the ambiguity in this scientific field. In the past various manual and physiotherapeutic exercise methods have already been tested.

This study is also intended to examine the effectiveness of muscle training for the treatment of patients with anterior disc displacement with reduction. The exercises are primarily supposed to train the lateral pterygoid muscle. The treatment with an equilibration appliance in the lower jaw serves as a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Orofacial pain in the joint or muscles, degree NRS≥3
* Clicking phenomenon during TMJ opening or closing movement
* Deviation movement during opening of the lower jaw
* Legal competence and presence of the signed declaration of consent

Exclusion Criteria:

* Drug abuse
* Depression
* Polyarthritis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
change orofacial pain: numeric rating scale (NRS; 0-10) | 2 months, 4 months, 6 months
  The primary outcome variable is defined as the change of orofacial pain in the head and joint area after initiating the therapy measured by numeric rating scale (NRS; 0-10, 0: no pain, 10: worst imaginable pain) at the time of the follow-up appointments

SECONDARY OUTCOMES:
Change in number of clicking noises | 2 months, 4 months, 6 months
  Change in number of clicking noises in the TMJ during jaw opening or jaw closing movements established by palpation of the TMJs
Change in interincisal distance during jaw opening | 2 months, 4 months, 6 months
  Change in interincisal distance during maximum unassisted opening measured in mm between first upper and lower right incisor. If one of the teeth is missing: first upper and lower left incisor
Change in force degrees for the lateral movement of the mandible (scale 0-5) | 2 months, 4 months, 6 months
  Evaluation of muscle forces during lateral jaw movements on a ordinal scale (0-5) according to Janda

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Bernhardt, Prof., Principal Investigator — University Medicine Greifswald
Locations (1):
- Zahnarztpraxis Dr. Pfanne, Steina, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bumann, A., Groot Landeweer, G.: Manuelle Untersuchungstechniken zur Manuellen Untersuchungstechniken zur Differenzierung von Funktionsstörungen im Kausystem. In Hahn, W.: Funktionslehre: aktueller Stand und praxisgerechte Umsetzung. Hanser, München, 1993
- [Background] Eberhard D, Bantleon HP, Steger W. The efficacy of anterior repositioning splint therapy studied by magnetic resonance imaging. Eur J Orthod. 2002 Aug;24(4):343-52. doi: 10.1093/ejo/24.4.343. PMID 12198864
- [Background] Egermark I, Magnusson T, Carlsson GE. A 20-year follow-up of signs and symptoms of temporomandibular disorders and malocclusions in subjects with and without orthodontic treatment in childhood. Angle Orthod. 2003 Apr;73(2):109-15. doi: 10.1043/0003-3219(2003)732.0.CO;2. PMID 12725365
- [Background] El-Asfahani I, Kortam S (2020) Effect of CAD/CAM versus conventional anterior repositioning splints on the management of temporomandibular joint disc displacement with reduction: A randomized controlled clinical trial. Egyptian Dental Journal 66:571-585. doi: 10.21608/edj.2020.79131
- [Background] Janda V (2013) Muscle Function Testing. Butterworth-Heinemann
- [Background] Kalaykova SI, Lobbezoo F, Naeije M. Risk factors for anterior disc displacement with reduction and intermittent locking in adolescents. J Orofac Pain. 2011 Spring;25(2):153-60. PMID 21528122
- [Background] Karacayli U, Mumcu G, Cimilli H, Sisman N, Sur H, Gunaydin Y. The effects of chronic pain on oral health related quality of life in patients with anterior disc displacement with reduction. Community Dent Health. 2011 Sep;28(3):211-5. PMID 21916356
- [Background] Kumazaki Y, Kawakami S, Hirata A, Oki K, Minagi S. Ipsilateral Molar Clenching Induces Less Pain and Discomfort than Contralateral Molar Clenching in Patients with Unilateral Anterior Disc Displacement of the Temporomandibular Joint. J Oral Facial Pain Headache. 2016 Summer;30(3):241-8. doi: 10.11607/ofph.1405. PMID 27472527
- [Background] Lindfors E, Arima T, Baad-Hansen L, Bakke M, De Laat A, Giannakopoulos NN, Glaros A, Guimaraes AS, Johansson A, Le Bell Y, Lobbezoo F, Michelotti A, Muller F, Ohrbach R, Wanman A, Magnusson T, Ernberg M. Jaw Exercises in the Treatment of Temporomandibular Disorders-An International Modified Delphi Study. J Oral Facial Pain Headache. 2019 Fall;33(4):389-398. doi: 10.11607/ofph.2359. Epub 2019 Jun 24. PMID 31247061
- [Background] List T, Axelsson S. Management of TMD: evidence from systematic reviews and meta-analyses. J Oral Rehabil. 2010 May;37(6):430-51. doi: 10.1111/j.1365-2842.2010.02089.x. Epub 2010 Apr 20. PMID 20438615
- [Background] McNeely ML, Armijo Olivo S, Magee DJ. A systematic review of the effectiveness of physical therapy interventions for temporomandibular disorders. Phys Ther. 2006 May;86(5):710-25. PMID 16649894
- [Background] Nagata K, Hori S, Mizuhashi R, Yokoe T, Atsumi Y, Nagai W, Goto M. Efficacy of mandibular manipulation technique for temporomandibular disorders patients with mouth opening limitation: a randomized controlled trial for comparison with improved multimodal therapy. J Prosthodont Res. 2019 Apr;63(2):202-209. doi: 10.1016/j.jpor.2018.11.010. Epub 2018 Dec 15. PMID 30563758
- [Background] Navi F, Kalantar Motamedi MH, Taheri Talesh K, Lasemi E, Nematollahi Z (2013) Diagnosis and Management of Temporomandibular Disorders. In: Kalantar Motamedi MH (ed) A Textbook of Advanced Oral and Maxillofacial Surgery. InTech
- [Background] Navi F, Motamedi MHK, TaheriTalesh K, Lasemi E, Nematollahi Z (2013) Diagnosis and Management of Temporomandibular Disorders. A Textbook of Advanced Oral and Maxillofacial Surgery. doi: 10.5772/55018
- [Background] Okeson JP. Long-term treatment of disk-interference disorders of the temporomandibular joint with anterior repositioning occlusal splints. J Prosthet Dent. 1988 Nov;60(5):611-6. doi: 10.1016/0022-3913(88)90224-7. PMID 3199322
- [Background] Okeson JP (2019) Management of Temporomandibular Disorders and Occlusion - E-Book. Elsevier Health Sciences
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Wanman A, Marklund S. Treatment outcome of supervised exercise, home exercise and bite splint therapy, respectively, in patients with symptomatic disc displacement with reduction: A randomised clinical trial. J Oral Rehabil. 2020 Feb;47(2):143-149. doi: 10.1111/joor.12888. Epub 2019 Sep 30. PMID 31520538
- [Background] Wieckiewicz M, Grychowska N, Wojciechowski K, Pelc A, Augustyniak M, Sleboda A, Zietek M. Prevalence and correlation between TMD based on RDC/TMD diagnoses, oral parafunctions and psychoemotional stress in Polish university students. Biomed Res Int. 2014;2014:472346. doi: 10.1155/2014/472346. Epub 2014 Jul 9. PMID 25121100
- [Background] Wolfart S, Heydecke G, Luthardt RG, Marre B, Freesmeyer WB, Stark H, Wostmann B, Mundt T, Pospiech P, Jahn F, Gitt I, Schadler M, Aggstaller H, Talebpur F, Busche E, Bell M. Effects of prosthetic treatment for shortened dental arches on oral health-related quality of life, self-reports of pain and jaw disability: results from the pilot-phase of a randomized multicentre trial. J Oral Rehabil. 2005 Nov;32(11):815-22. doi: 10.1111/j.1365-2842.2005.01522.x. PMID 16202045
- [Background] Wright EF, Klasser GD (2019) Manual of Temporomandibular Disorders. John Wiley & Sons
- [Background] Wright EF, North SL. Management and treatment of temporomandibular disorders: a clinical perspective. J Man Manip Ther. 2009;17(4):247-54. doi: 10.1179/106698109791352184. PMID 20140156

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04819763/Prot_SAP_000.pdf